CLINICAL TRIAL: NCT06257368
Title: TFL-DUST Study TFL Driven Urinary System Treatment Study
Brief Title: TFL Driven Urinary System Treatment Study
Acronym: TFL-DUST
Status: Recruiting | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CP359
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Urologic Diseases
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Coloplast TFL Drive — Thulium Fiber laser

SUMMARY:
The goal of this observational study is:

To assess the use of Coloplast TFL Drive in daily practice

To confirm:

* the safety and efficacy of the Coloplast TFL Drive and its GUI (Graphical User Interface) with pre-embedded settings in Laser lithotripsy
* the safety and efficacy of the Coloplast TFL Drive and its GUI with pre-embedded settings for enucleation of prostate as treatment of benign prostate hyperplasia
* the safety and efficacy of the Coloplast TFL Drive and its GUI with pre-embedded settings for ablation of urological tumors

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient, for which TFL laser is indicated for treating a urological disease (e.g. kidney or ureteral stones, urological tumor, BPH (Benign Prostate Hypertrophy…)

Exclusion Criteria:

* Any condition when TFL laser should not be indicated as per the TFL user manual (untrained surgeon on laser use, patient's conditions)
* Patients with no signed consent form
* Patients <18 years old
* Patients under tutorship or guardianship
* Patients who already took part in the study
* Pregnant or breastfeeding women
* Patient undergoing 2nd step laser procedure at inclusion
* Subject already included in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients, male and female with an urological disease for which TFL treatment is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time in Laser ON | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle D de Berny, Study Director — Coloplast Manufacturing France
Locations (5):
- France (4):
  - CHU Bordeaux, Bordeaux
  - Clinique Jules Verne, Nantes
  - Hôpital Tenon, Paris
  - Hôpital Privé Francheville, Périgueux
- HM Hospital Sanchinarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No